CLINICAL TRIAL: NCT04928105
Title: Clinical Study of Senl-T7 CAR-T Cells in the Treatment of Relapsed or Refractory CD7+ Lymphoma
Brief Title: Senl-T7 CAR-T Cells for Treatment of Relapsed or Refractory CD7+ Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Senl-T7 CART for CD7+ lymphoma
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2021-06

CONDITIONS: Lymphoma, T-Cell
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD7 CAR-T (Experimental)
  Interventions: Biological: Senl-T7

INTERVENTIONS:
Biological: Senl-T7 — Patients will be treated with CD7 CAR-T cells

SUMMARY:
This study is an open and prospective clinical study, taking patients with relapsed or refractory CD7+ lymphoma as the test subjects, in order to evaluate the safety and efficacy of Senl-T7 CAR-T for patients with CD7+ lymphoma.

DETAILED DESCRIPTION:
Main research purposes:

To evaluate the safety and efficacy of Senl-T7 CAR-T for relapsed or refractory CD7+ lymphoma

Secondary research purpose:

To investigate the cytokinetic characteristics of Senl-T7 CAR-T for relapsed or refractory CD7+ lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed as relapsed or refractory lymphoma; 2. Tumor cells express CD7 (express CD7 by flow cytometry or immunohistochemistry); 3. The expected survival period is greater than 12 weeks; 4. KPS or Lansky score ≥60; 11 5. Age 2-70 years old; 6. HGB≥70g/L (can be transfused); 7. Indoor blood oxygen saturation> 90%; 8. Total bilirubin does not exceed 3 times the upper limit of normal value, and AST and ALT do not exceed 5 times the upper limit of normal value; 9. The subject or guardian understands and signs the informed consent form;

Exclusion Criteria:

* 1. One of the following cardiac criteria: atrial fibrillation; myocardial infarction within the past 12 months; prolonged QT synthesis Syndrome or secondary QT prolongation is at the discretion of the investigator. Echocardiography LVSF<30% or LVEF< 50%; clinically significant pericardial effusion; cardiac insufficiency NYHA (New York Heart Association) III or IV (the absence of this symptom confirmed by echocardiography within 12 months after treatment); 2. There is active GVHD; 3. Have a history of severe pulmonary dysfunction diseases; 4. Merge other malignant tumors in advanced stage; 5. Combined with severe infection or persistent infection and cannot be effectively controlled; 6. Combined with severe autoimmune disease or congenital immunodeficiency; 7. Active hepatitis (hepatitis B virus deoxyribonucleic acid [HBVDNA] or hepatitis C virus ribonucleic acid [HCVRNA] test positive); 8. Human immunodeficiency virus (HIV) infection or syphilis infection or HTLV infection; 9. There is a history of severe allergies to biological products (including antibiotics); 10. Clinically significant viral infection, or uncontrollable viral reactivation, including EBV (Epstein-Barr virus), CMV (cytomegalovirus), ADV (adenovirus), BKV, HHV(human herpesvirus)-6; 11. There are central nervous system disorders, such as uncontrolled epilepsy, cerebrovascular ischemia/hemorrhage, dementia, Cerebellar diseases, etc.; 12. Female patients are pregnant and lactating, or have a pregnancy plan within 12 months; 13. Circumstances that the researcher believes may increase the risk of the subject or interfere with the results of the test.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First 1 month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after CD7
Remission Rate | 3 months post CAR-T cells infusion
  Remission Rate including complete remission(CR)、CR with incomplete blood count recovery(CRi)、No remission(NR)
duration of response (DOR) | 24 months post CAR-T cells infusion
  duration of response (DOR)
progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of CD7 CAR- T cells in the genomes of PBMC by qPCR method
CAR-T proliferation | 3 months post CAR-T cells infusion
  percentage of CD7 CAR- T cells measured by flow cytometry method
Cytokine release | First 1 month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry method

CONTACTS AND LOCATIONS:
Overall Officials: Peihua MD Lu, PhD, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei yanda Ludaopei Hospital, Yanda, Hebei, China